CLINICAL TRIAL: NCT06331715
Title: An Open Label, Balanced, Randomized, Two Treatments, Two Sequences, Two Periods, Single Dose, Crossover Bioequivalence Study of Palbociclib 125 mg Capsules (Iclos) and Ibrance (Palbociclib) 125 mg Capsules Pfizer in Healthy Subjects Under Fed Condition
Brief Title: Bioequivalence Study of Palbociclib 125 mg Capsules of Iclos vs. Ibrance (Palbociclib) Capsules 125 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Megalabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ML1005
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Bioequivalence
Keywords: palbociclib
MeSH Terms: interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR (Experimental): Subject will receive Test product palbociclib (125 mg Iclos) followed by reference product (Ibrance Pfizer 125 mg capsules) after 14 days washout
  Interventions: Drug: Palbociclib 125mg
- RT (Experimental): Subject will receive reference product (Ibrance Pfizer 125 mg capsules) followed by Test product palbociclib (125 mg Iclos) after 14 days washout
  Interventions: Drug: Palbociclib 125mg

INTERVENTIONS:
Drug: Palbociclib 125mg — Pharmacokinetic parameters AUC and Cmax will be evaluated to establish bioequivalence betweeen the Test and Reference products
  Other Names: Ibrance; Palbociclib Iclos

SUMMARY:
An open label, balanced, randomized, two treatments, two sequences, two periods, cross over, single dose, bioequivalence study of Palbociclib 125 mg Capsules of Iclos Uruguay S.A and IBRANCE® (Palbociclib) 125 mg Capsules of Pfizer Europe (Belgium) in healthy, adult, human subjects under fed condition.

DETAILED DESCRIPTION:
24 healthy subjects males and/or non pregnant, non breast feeding females will be randomized to receive either Test product (Palbociclib 125 mg Capsules of Iclos Uruguay S.A.) or Reference product (Ibrance® Palbociclib 125 mg Capsules of Pfizer Europe in healthy, adult, human subjects under fed condition. Trial design will be balanced, randomized, two treatments, two sequences, two periods, cross over, single dose, bioequivalence study of in healthy, adult, human subjects under fed condition to assess the bioequivalence between test and comparator formulations.

Statistical analysis will be performed on the Ln-transformed pharmacokinetic parameters using SAS® v 9.4. The analysis will include data from subjects who complete the study. If there are dropouts, no replacement will be done.

To establish bioequivalence of the test product with that of comparator product, 90% Confidence Interval (CI) for the ratio (Test/ Comparator) of Least Square Means of the log transformed PK parameters (Cmax and AUC0-72) must fall between 80.00% and 125.00%. Confidence Interval (CI) values will not be rounded off.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or non-pregnant, non-breast feeding female literate volunteers of 18 to 45 years (both years inclusive) with BMI of 18.50 - 30.00 Kg/m2 and weight > 50 Kg.
* Healthy volunteers as evaluated by medical history, vitals and general clinical examination.
* Normal or clinically insignificant biochemical, hematological, urine and serology parameters.
* Normal or clinically insignificant ECG.
* Negative urine test for drugs of abuse and alcohol breath analysis for both males and females,
* Negative pregnancy test for females and do not plan to become pregnant during course of the study and for 03 months after completion of study.
* Volunteers who are willing to use acceptable methods of contraception during course of the study and for 03 months after completion of study.
* Volunteers who can give voluntary written informed consent and communicate effectively.

Exclusion Criteria:

* History of any major surgical procedure in the past 03 months.
* History of any clinically significant cardiac, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric and hematological disorders.
* History of chronic alcoholism/ chronic smoking/ drug of abuse.
* Volunteers with known hypersensitivity to Palbociclib or any of the excipients.
* History of consumption of tobacco containing products within 48 hours prior to proposed time of dosing
* Volunteer who are positive for hepatitis B surface antigen, anti-hepatitis C antibody, treponemal antibodies and human immunodeficiency virus (HIV 1&2) antibodies.
* Present or past history of intake of drugs or any prescription drug or over the counter (OTC) drugs/ vaccines (including COVID 19 vaccines) within 14 days which potentially modify kinetics / dynamics of Palbociclib or any other medication judged to be clinically significant by the investigator.
* History of consumption of grapefruit and/or its products within 10 days prior to the start of study.
* Volunteer who had participated in any other clinical study or who had bled during the last 03 months before check-in.
* History of consumption of one or more of the below, 48 hours prior to dosing:

Xanthine containing food or drinks such as cola, chocolate, coffee or tea, citrus fruits or items (lime, lemon and orange), alcohol and any other food/beverage known to have interactions as deemed by the investigator

* History of difficulties in swallowing tablets/capsules.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
AUC 0-t | 72 hours
  Least Square Means of Test/Reference Ratio of Area Under Plasma concentration vs. time between 80-125 for 90%IC
Cmax | 72 hours
  Least Square Means of Test/Reference Ratio of maximum plasma concentration between 80-125 for 90%IC

CONTACTS AND LOCATIONS:
Overall Officials: M Gowtham, MD, Principal Investigator — Azidus Laboratories
Locations (1):
- Azidus Laboratories, Chennai, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA guidance for the bioequivalence of dasatinib — https://www.accessdata.fda.gov/drugsatfda_docs/psg/PSG_212436.pdf
- See also: EMA bioequivalence guideline for palbociclib — https://www.ema.europa.eu/en/documents/scientific-guideline/palbociclib-hard-capsule-75-mg-100-mg-and-125-mg-and-film-coated-tablet-75-mg-100-mg-and-125-mg-product-specific-bioequivalence-guidance-revision-1_en.pdf